CLINICAL TRIAL: NCT05786976
Title: Assessment of Skin Tolerance and Efficacy of a Cosmetic Product After 4 Weeks of Use on Subjects With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CSBL01-ICBD
Record Dates: First submitted 2023-02-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Atopic Diathesis; Eczema-Prone Skin

STUDY DESIGN:
Intervention Model Description: intra-individual comparison
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lotion BNO 3732 for topical care (Experimental)
  Interventions: Other: Lotion BNO 3732
- Body Lotion Benchmark product for topical care (Active Comparator)
  Interventions: Other: Body Lotion Benchmark product

INTERVENTIONS:
Other: Lotion BNO 3732 — Crem body lotion twice daily
  Arms: Lotion BNO 3732 for topical care
Other: Body Lotion Benchmark product — Crem body lotion twice daily
  Arms: Body Lotion Benchmark product for topical care

SUMMARY:
The aim of this study is to compare the efficacy and tolerability of a cosmetic product to one that is already available on the market (benchmark product). Efficacy is assessed by instrumental measurements of skin condition, clinical examinations, and questionnaires.

DETAILED DESCRIPTION:
The objective of this exploratory study is to investigate the efficacy and tolerability of a cosmetic product on subjects with atopic dermatitis after 4 weeks of use in comparison to a benchmark product.

The efficacy will be evaluated via instrumental measurements of skin hydration by Corneometer, transepidermal water loss by Tewameter and erythema by Chromameter. Furthermore, the efficacy was evaluated by dermatological assessment using the local SCORing Atopic Dermatitis (SCORAD) rated by a dermatologist in the children, the dermatological assessment rated by a dermatologist (objective) and the dermatological assessment rated by adult subject (subjective) in the test areas, respectively.

Additionally, at the beginning and at the end of the study the Patient-Oriented Eczema Measure (POEM) will be evaluated by the subjects or the subjects' parents/legal guardians by questionnaires.

The SCORAD evaluation and the objective and subjective dermatological assessments will also be used for the tolerability assessment of the test products.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the subject to participate in the study, or, for underage subjects of the parents/ legal guardians to let their child participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits or, for underage subjects, willingness of the parents/ legal guardians to actively support their child's participation in the study and to come to the scheduled visits with their child
* Female and/or male
* Children from 6 months to 14 years of age and adults between 18 and 65 years of age
* Eczema-prone skin and atopic diathesis, diagnosed by the dermatologist

Exclusion Criteria:

* Female subjects: pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* Insulin-dependent diabetes mellitus
* One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension, cardiovascular diseases
* Documented allergies to cosmetic products and/ or ingredients, skin care and/or skin cleansing products
* Wounds, moles, tattoos, scars, excessive hair growth, etc. at the test area that could influence the investigation
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. antiallergics) within the last 7 days prior to the start of the study
* Systemic therapy with anti-phlogistic agents or analgetics (e.g. diclophenac), except for minor pain relief medicine like acetylsalicylic acid or paracetamol within the last 3 days prior to the start of the study

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in transepidermal water loss (g/m2h) | 29 days
Mean change from baseline in skin redness by Chromameter | 29 days
Mean change from baseline in skin hydration (Skin capacitance by Corneometer [a.u.]) | 29 days
Changes from baseline in local SCORAD (Scoring Atopic Dermatitis, min=0, max=3; 3=worse outcome) in children | 29 days
Changes from baseline in objective dermatological evaluation of skin status (erythema, dryness, scaling, fissures, papules, pustules, edema, vesicles, weeping) by dermatologist | 29 days
Changes from baseline in POEM (Patient-oriented eczema measure, min=0, max=28; 28=worse outcome) | 29 days

SECONDARY OUTCOMES:
Change from baseline in the scoring of subjective dermatological evaluation via questionnaire (adults) (min=0, max=3; 3=worse outcome) | 29 days
Evaluation of products traits via questionnaire (20 questions with different answers, no scales) | Day 1, after first application
Evaluation of products traits via questionnaire (20 questions with different answers, no scales) | 8 days
Evaluation of products traits via questionnaire (20 questions with different answers, no scales) | 29 days
Safety of BNO 3732 measured by reported Adverse Events | until day 29

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Laing, Dr., Principal Investigator — proDERM GmbH
Locations (1):
- SGS proderm GmbH, Schenefeld, Germany